CLINICAL TRIAL: NCT06398964
Title: Effects of 2-week Ketosis on Myocardial Ketone Body Consumption, Utilization, and External Efficiency in Patients With Chronic Heart Failure
Brief Title: Effects of 2-week Ketosis on the Heart's Ketone Body Consumption, Utilization, and Energetic Efficiency in Patients With Chronic Heart Failure
Acronym: KETO-CHF PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Wiggers, Professor, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: KETO-CHF-PET
Record Dates: First submitted 2023-08-23; First posted 2024-05-03 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3-hydroxybutyrate (Active Comparator)
  Interventions: Dietary Supplement: 3-hydroxybutyrat
- Isocaloric placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Isocaloric placebo drink

INTERVENTIONS:
Dietary Supplement: 3-hydroxybutyrat — The intervention is administered as a drink.
  Arms: 3-hydroxybutyrate
Dietary Supplement: Isocaloric placebo drink — The intervention is administered as a drink.
  Arms: Isocaloric placebo drink

SUMMARY:
Heart Failure (HF) is a significant health concern, affecting around 1-2% of people in Western countries. The risk of developing HF during a lifetime is about 20%. Despite advancements in HF care, the one-year mortality rate for HF patients remains high. HF patients also experience reduced physical capacity and quality of life. The heart relies heavily on a process called oxidative metabolism for energy, and this process requires a continuous supply of energy sources like fatty acids, glucose, and ketone bodies. In HF, there's a shift in how the heart uses these energy sources, which affects its efficiency.

Ketone bodies such as 3-OHB, are molecules that can provide the heart with a more efficient energy source compared to traditional ones like fatty acids or glucose. They are produced in the liver and are important for supplying energy during fasting, exercise, and illness. Recent research suggests that 3-OHB might have benefits for HF patients beyond just providing energy. It seems to reduce inflammation and oxidative stress in the heart. Some studies in healthy individuals have shown that infusing 3-OHB increases blood flow to the heart.

In HF patients, the investigators aim to explore the cardiac effects of a two-week supplement of 3-OHB. The aim is to investigate if this supplement can increase the heart's consumption and utilization of 3-OHB. The study involves 12 patients with HF and reduced ejection fraction (HFrEF). The patients will receive a ketone ester supplement four times a day for two weeks, and then they'll take an isocaloric placebo supplement for another two weeks.

The investigators will use positron emission tomography (PET) to study the cardiac oxygen consumption and 3-OHB uptake. This is done by injection of tracers (11-C-3-OHB and 11-C-acetate).

The study will also look at myocardial external efficiency (MEE) and myocardial blood flow (MBF). For a subset of participants, the investigators will also take myocardial biopsies and perform more detailed analyses, e.g. respirometry and electron microscopy or single nucleus mRNA sequencing, proteomics and metabolimcs, to understand the impact of the supplement on the heart's cellular structures and functions, transcriptome, proteome and metabolome.

Ultimately, this study aims to determine whether supplementing HF patients with 3-OHB can improve the heart's energy usage and potentially provide other beneficial effects. This research might pave the way for new treatments that enhance the heart's function and quality of life for HF patients.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes or HbA1c > 48 mmol/L
* significant cardiac valve disease
* severe stable angina pectoris
* severe comorbidity as judged by the investigator
* inability to give informed consent
* Age <55 years
* Other disease or treatment making subject unsuitable for study participation as judged by the investigator

Exclusion Criteria:

* Chronic heart failure
* NYHA class II-III
* left ventricular ejection fraction (LVEF) <40%
* Negative urine-HCG for women with childbearing potential

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Myocardial consumption of 3-OHB. | Participants meet for 2 examination days 4 weeks apart. This is a whole day involving 4 PET/CT scans each day.
  Uptake of the ketone radiotracer measured in µmol/min/g tissue in the myocardium will be calculated using kinetic modeling techniques using aQuant Research software.

SECONDARY OUTCOMES:
Myocardial oxygen consumption (MVO2) | Participants meet for 2 examination days 4 weeks apart. This is a whole day involving 4 PET/CT scans each day.
  Uptake and oxidation of the acetate radiotracer measured in mL/g/min tissue in the myocardium will be calculated using kinetic modeling techniques using aQuant Research software
Myocardial external efficacy | Participants meet for 2 examination days 4 weeks apart. This is a whole day involving 4 PET/CT scans each day.
  Refers to a measure that assesses how effectively the heart converts its energy consumption into external work. It's a parameter that evaluates the efficiency of the heart's mechanical function in relation to its energy utilization.
High resolution respirometry | Participants meet for 2 examination days 4 weeks apart. For a subset of participants, 1 myocardial biopsy and 2 skeletal muscle biopsies will be taken at each examination day.
  Picomolar/second/mg tissue. This unit quantifies the rate at which oxygen is consumed by the biological sample being studied.
Single nucleus mRNA sequencing of skeletal muscle and cardiomyocytes. | Participants meet for 2 examination days 4 weeks apart. For a subset of participants, 1 myocardial biopsy and 2 skeletal muscle biopsies will be taken at each examination day.
  Sequencing of mRNA (the transcriptome) from the nucleus of a single skeletal muscle cell and cardiomyocyte.
Proteomics of skeletal muscle and myocardial biopsies. | Participants meet for 2 examination days 4 weeks apart. For a subset of participants, 1 myocardial biopsy and 2 skeletal muscle biopsies will be taken at each examination day.
  Systematic analysis of the entire complement of proteins (the proteome) present in the skeletal muscle and myocardial biopsies. This includes identifying proteins, determining their abundance, studying their post-translational modifications.
Metabolomics of skeletal muscle and myocardial biopsies. | Participants meet for 2 examination days 4 weeks apart. For a subset of participants, 1 myocardial biopsy and 2 skeletal muscle biopsies will be taken at each examination day.
  Characterizing the entire complement of metabolites (the metabolome) in the skeletal muscle and myocardial biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Henrik, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savarese G, Lund LH. Global Public Health Burden of Heart Failure. Card Fail Rev. 2017 Apr;3(1):7-11. doi: 10.15420/cfr.2016:25:2. PMID 28785469
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Kolwicz SC Jr, Purohit S, Tian R. Cardiac metabolism and its interactions with contraction, growth, and survival of cardiomyocytes. Circ Res. 2013 Aug 16;113(5):603-16. doi: 10.1161/CIRCRESAHA.113.302095. PMID 23948585
- [Background] Selvaraj S, Kelly DP, Margulies KB. Implications of Altered Ketone Metabolism and Therapeutic Ketosis in Heart Failure. Circulation. 2020 Jun 2;141(22):1800-1812. doi: 10.1161/CIRCULATIONAHA.119.045033. Epub 2020 Jun 1. PMID 32479196
- [Background] Gormsen LC, Svart M, Thomsen HH, Sondergaard E, Vendelbo MH, Christensen N, Tolbod LP, Harms HJ, Nielsen R, Wiggers H, Jessen N, Hansen J, Botker HE, Moller N. Ketone Body Infusion With 3-Hydroxybutyrate Reduces Myocardial Glucose Uptake and Increases Blood Flow in Humans: A Positron Emission Tomography Study. J Am Heart Assoc. 2017 Feb 27;6(3):e005066. doi: 10.1161/JAHA.116.005066. PMID 28242634
- [Background] Yurista SR, Nguyen CT, Rosenzweig A, de Boer RA, Westenbrink BD. Ketone bodies for the failing heart: fuels that can fix the engine? Trends Endocrinol Metab. 2021 Oct;32(10):814-826. doi: 10.1016/j.tem.2021.07.006. Epub 2021 Aug 26. PMID 34456121
- [Background] Nielsen R, Moller N, Gormsen LC, Tolbod LP, Hansson NH, Sorensen J, Harms HJ, Frokiaer J, Eiskjaer H, Jespersen NR, Mellemkjaer S, Lassen TR, Pryds K, Botker HE, Wiggers H. Cardiovascular Effects of Treatment With the Ketone Body 3-Hydroxybutyrate in Chronic Heart Failure Patients. Circulation. 2019 Apr 30;139(18):2129-2141. doi: 10.1161/CIRCULATIONAHA.118.036459. PMID 30884964
- [Background] Monzo L, Sedlacek K, Hromanikova K, Tomanova L, Borlaug BA, Jabor A, Kautzner J, Melenovsky V. Myocardial ketone body utilization in patients with heart failure: The impact of oral ketone ester. Metabolism. 2021 Feb;115:154452. doi: 10.1016/j.metabol.2020.154452. Epub 2020 Nov 26. PMID 33248064
- [Background] Ho KL, Zhang L, Wagg C, Al Batran R, Gopal K, Levasseur J, Leone T, Dyck JRB, Ussher JR, Muoio DM, Kelly DP, Lopaschuk GD. Increased ketone body oxidation provides additional energy for the failing heart without improving cardiac efficiency. Cardiovasc Res. 2019 Sep 1;115(11):1606-1616. doi: 10.1093/cvr/cvz045. PMID 30778524
- [Background] Thai PN, Miller CV, King MT, Schaefer S, Veech RL, Chiamvimonvat N, Bers DM, Dedkova EN. Ketone Ester D-beta-Hydroxybutyrate-(R)-1,3 Butanediol Prevents Decline in Cardiac Function in Type 2 Diabetic Mice. J Am Heart Assoc. 2021 Oct 5;10(19):e020729. doi: 10.1161/JAHA.120.020729. Epub 2021 Sep 29. PMID 34583524